CLINICAL TRIAL: NCT05594706
Title: Anhydroglucitol as a Measure of the Functional Beta-cell Mass in Children With Type 1 Diabetes - Pilot Study
Brief Title: Anhydroglucitol in Children With Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Philippe Klee, MD-PhD, Principal investigator, University Hospital, Geneva
Other Study IDs: 2022-01684
Record Dates: First submitted 2022-09-29; First posted 2022-10-26 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Newly diagnosed patients with T1DM: The investigators will do prospective measures in 10 to 15 children aged 2 to 18 years, at the time of diagnosis, four months after diagnosis and one year after diagnosis.
  Interventions: Other: Measurement of blood levels of 1,5-anhydroglucitol
- Patients with T1DM of different duration: As the functional beta-cell mass gradually declines as disease duration increases, the investigators will do measurements in a cohort of children aged ≤ 18 years, with increasing diabetes duration. The investigators plan to analyze groups of 5 patients with a disease duration of 3 (36 - 47 months), 5 (60 - 71 months) and 10 years (120 - 131 months), respectively.
  Interventions: Other: Measurement of blood levels of 1,5-anhydroglucitol

INTERVENTIONS:
Other: Measurement of blood levels of 1,5-anhydroglucitol — Measurement of blood levels of 1,5-anhydroglucitol

SUMMARY:
The investigators will measure blood levels of 1,5-anhydroglucitol in children with type 1 diabetes and correlate them with parameters related to functional beta-cell mass in diabetic patients. The values will be compared to those obtained in healthy volunteers. Children with newly diagnosed diabetes as well as children with longstanding disease will be included. The aim of the study is to test the validity of 1,5-anhydroglucitol as a novel biomarker of beta-cell mass and function in type 1 diabetes.

DETAILED DESCRIPTION:
One-center prospective exploratory pilot study performed in collaboration between the Pediatric Endocrine and Diabetology unit of the University Hospitals of Geneva (HUG) and Prof. Pierre Maechler, Diabetes Center of the Faculty of Medicine, University of Geneva Switzerland.

1,5-anhydroglucitol (1,5-AG), a deoxyhexose present in almost all foods and forming a stable pool in human subjects, has recently been found to be correlated with functional beta-cell mass in two different mouse models of beta-cell dysfunction leading to diabetes. The decline of this biomarker precedes the development of hyperglycemia in lean b-Phb2 -/- and obese db/db diabetic mice, where beta-cell loss occurs through two different mechanisms.

Additional studies have shown a correlation of 1,5-AG levels with risk of progression of type 1 diabetes (T1DM) in auto-antibody positive children, as well as with glycaemic control in patients with type 2 diabetes.

The present project will analyse the correlation between functional beta-cell mass and the circulating levels of 1,5-AG in children with T1DM. This should contribute to the evaluation of a novel biomarker of beta-cell mass and function in T1DM.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes with positive autoantibodies against islets, insulin, islet antigen 2 (IA2), glutamic acid decarboxylase (GAD) 65 or zinc transporter (ZnT)8.
* Treatment with continuous subcutaneous insulin infusion (CSII) with or without automated insulin delivery (AID).
* Monitoring with a continuous glucose measurement system (CGMS) or flash glucose monitor (FGM).
* Patient willing to keep the same type of CGMS or FGM during the year of observation
* Ability to give informed consent as documented by signature

Exclusion Criteria:

* Patients treated with multiple daily injections (MDI) or not willing to wear a CGMS of FGM
* Patients changing the type of CGMS during the course of the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Among children with type 1 diabetes, aged 2 to 18 years:
  15 newly diagnosed patients and 15 age- and sex-matched controls. 5 patients with a diabetes duration of 3 (36 - 47 months), 5 patients with a disease duration of 5 (60 - 71 months) and 5 patients with a disease duration of 10 years (120 - 131 months) and 15 corresponding age- and sex-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of 1,5-anhydroglucitol levels in newly diagnosed patients with indirect markers of beta-cell function and mass | Day 1
  Blood levels of 1,5-anhydroglucitol will be correlated with indirect markers of beta-cell function at different moments after diagnosis
Correlation of 1,5-anhydroglucitol levels in newly diagnosed patients with indirect markers of beta-cell function and mass | 4 months after diagnosis
  Blood levels of 1,5-anhydroglucitol will be correlated with indirect markers of beta-cell function at different moments after diagnosis
Correlation of 1,5-anhydroglucitol levels in newly diagnosed patients with indirect markers of beta-cell function and mass | 12 months after diagnosis
  Blood levels of 1,5-anhydroglucitol will be correlated with indirect markers of beta-cell function at different moments after diagnosis
Correlation of 1,5-anhydroglucitol levels in patients with longstanding disease with indirect markers of beta-cell function and mass | In participants with a disease duration of 3 years.
  Blood levels of 1,5-anhydroglucitol will be correlated with indirect markers of beta-cell function in patients with different disease duration
Correlation of 1,5-anhydroglucitol levels in patients with longstanding disease with indirect markers of beta-cell function and mass | In participants with a disease duration of 5 years.
  Blood levels of 1,5-anhydroglucitol will be correlated with indirect markers of beta-cell function in patients with different disease duration
Correlation of 1,5-anhydroglucitol levels in patients with longstanding disease with indirect markers of beta-cell function and mass | In participants with a disease duration of 10 years.
  Blood levels of 1,5-anhydroglucitol will be correlated with indirect markers of beta-cell function in patients with different disease duration

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided